CLINICAL TRIAL: NCT05643339
Title: The Reproducibility of Microvascular Flow in Fibroids and Its Correlation With 2D and 3D Power Doppler Outcomes: a Prospective Cohort Study
Brief Title: The Reproducibility of Microvascular Flow Imaging in Fibroids and Its Correlation With 2D and 3D Power Doppler Outcomes
Acronym: MVF
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Marjolein Spiering, Investigator Reseach Office Womens Child Center, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2017/494 and W20_274
Record Dates: First submitted 2022-11-01; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Fibroid Uterus
Keywords: fibroid; microvascular flow; power doppler
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: microvascular flow imaging — microvascular flow imaging

SUMMARY:
The investigators hypothesized that Macrovascular Flow imaging could contribute to 2D power Doppler and 3D power Doppler in depicting fibroid vascularity. However, data concerning the feasibility and reproducibility of Macrovascular Flow imaging is lacking. Therefore the purpose of our study was to determine 1) the reproducibility of Macrovascular Flow imaging, 2) its correlation with 2D and 3D power Doppler, and 3) penetration depth, in order to investigate the added value for daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* one or more uterine fibroids
* diameter between 1,5 and 12 cm
* fibroid easily recognizable on ultrasound

Exclusion Criteria:

* younger than 18 years
* pregnancy
* uterine or cervical malignancy
* adenomyosis.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Eligible patients were women with one or more uterine fibroids, with a diameter between 1,5 and 12 cm, of which one was easily recognizable on ultrasound to assure the quality of the Doppler images.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
reproducibility by inter- and intraobserver agreement | Day 1
  The primary outcome was calculated by the assessment of intercorrelation coefficient (ICC) and its 95% confidence interval (CI) using a two-way mixed model. An ICC value of 0.75-1.00 indicates a good to excellent agreement(19). Bland-Altman plots showed the distribution of data.

SECONDARY OUTCOMES:
penetration in centimeters | Day 1
  The penetration was measured along the direction of the ultrasound wave, from the probe to the deepest ultrasound signal visible, both for Microvascular Flow and power Doppler. Differences in ordinal data was tested by Mann Whitney U, non-normal continuous data by Wilcoxon rank test and normally distributed continuous data by a one sample t-test.
architecture | Day 1
  architecture of vessels visible in different regions yes/no.
presence doppler signal | Day 1
  yes/no in different regions

CONTACTS AND LOCATIONS:
Overall Officials: Judith Huirne, Prof., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No